CLINICAL TRIAL: NCT02863731
Title: Effect of Alternating Postures on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences Upper Austria (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Schwartz, Research Associate, University of Applied Sciences Upper Austria
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AO-8735-2; 834185 (Other Grant/Funding Number: Austrian Research Promotion Agency (FFG))
Record Dates: First submitted 2016-07-14; First posted 2016-08-11 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Sedentary Lifestyle
Keywords: postural changes; alternating postures; Cognitive performance; Height-adjustable desk; Worksite
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alternating postures: first day (Experimental): Alternating body postures on the first day of measurement. Sitting body posture on the second day of measurement.
  Interventions: Other: Alternating working postures, first day
- Alternating postures: second day (Experimental): Alternating body postures on the second day of measurement. Sitting body posture on the first day of measurement.
  Interventions: Other: Alternating working postures, second day
- Control group (No Intervention): Sitting body posture on both days of measurement.

INTERVENTIONS:
Other: Alternating working postures, first day — On the first day of measurement participants execute five test battery trials in alternating postures (sit/stand/sit/stand/sit). On the second day of measurement participants execute the test battery in a sitting posture (sit/sit/sit/sit/sit).
  Arms: Alternating postures: first day
Other: Alternating working postures, second day — On the first day of measurement participants execute five test battery trials in a sitting posture (sit/sit/sit/sit/sit). On the second day of measurement participants execute the test battery in alternating postures (sit/stand/sit/stand/sit).
  Arms: Alternating postures: second day

SUMMARY:
Prolonged sitting is a risk factor for cardiovascular and musculoskeletal diseases, diabetes, several types of cancer and all-cause mortality. In combination with static and awkward postures, the prevalence of musculoskeletal diseases can increase further. Although the implementation of sit-to-stand or active workstations can help to reduce sitting time, improve physical activity at work and promote health benefits, it might also lead to changes in cognitive functions such as productivity. The purpose of this study is to evaluate the short-term effect of alternating working postures on cognitive performance for healthy people.

DETAILED DESCRIPTION:
Measurements were made in a laboratory. They were made on two different days with an interval of 7 days between sessions. Laboratory tests were conducted in a controlled, simulated work-space located at the University of Applied Sciences Campus Linz. All laboratory measurements were made in a controlled laboratory at the campus site Linz of the University of Applied Sciences Upper Austria. Temperature, air flow, humidity, lighting conditions (artificial light only) and noise level were controlled and set to be consistent with the subjects' typical working environment.

During the laboratory measurements, subjects either stood or sat upright in an ergonomic office chair, according to the study protocol. Subjects were encouraged to work as fast and as accurately as they could. To ensure identical testing conditions between subjects and to not unduly influence physiological parameters such as heart rate variability (HRV), subjects were required to minimize excessive movement (e.g. standing up during the sitting periods).

In the first (initial) phase participants were familiarized with the study protocol. Sitting time and weekly physical activity were determined via the long version of the International Physical Activity Questionnaire (IPAQ, only on the first day of measurement). Examples of each cognitive test implemented in the cognitive phase were executed according to their guidelines. A 30 minute break in a sitting posture was used to ascertain baseline heart-rate level. Baseline heart-rate was calculated after a 20 minute rest for a 5 minute interval.

In the second (cognitive) phase subjects participated in a test battery containing five blocks. Each block consisted of a working speed test (text editing task), an attentional test (d2R-test of attention) and a reaction time test (Stroop-test). These tests lasted for 30 minutes to fulfill recommendations regarding postural changes. To simulate "common" working conditions (computer based and non-computer based tasks), digital (text editing task, Stroop-test) as well as pen & paper (d2R-test) versions of the implemented tests were used.

For the intervention group, the cognitive blocks were executed in an alternating posture (sit - stand - sit - stand - sit) either on the first or the second day of measurement (cross-over design). To generate control periods, this procedure was executed in an sitting posture only (sit - sit - sit - sit - sit) for the non-interventional day. For the control group, both days of measurement were executed in sitting posture only (sit - sit - sit - sit - sit ).

In the third (final) phase participants were asked to estimate their workload by means of the Task Load Index questionnaire developed by the National Aeronautics and Space Administration (NASA-TLX), followed by a 30 minutes resting phase in a sitting posture. During both 30 min resting phases (initial & final) participants watched documentaries and were encouraged not to talk.

Heart-rate and trunk movements were measured from the start of the study protocol until the next morning by means of an mobile ECG-recorder.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian (no acute or chronic diseases)
* Normal weight or overweight (BMI: 18.5 - 30.0 kg/m²)
* Regular computer users
* Fluent German speakers
* Consented to participate

Exclusion Criteria:

* Obesity (BMI > 30.0 kg/m²)
* Experience in sit-to-stand workstations
* Acute or chronic diseases
* Inability to stand
* Visual impairments that had not been corrected
* Color blindness
* Regular heavy smokers (> 10 cigarettes /day)
* Not consented to participate

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Reaction time | 2 experimental days
  Reaction time is a commonly measured parameter to describe mental states, fatigue or performance in ergonomic research. As the effect of alternating postures on reaction time is still unclear, a digital version of the Color-Word-Conflict-Stroop-Test has been implemented.
  It contained 190 congruent, incongruent and neutral tasks and required approximately 10 min to simulate long-lasting monotonous office screen work. The reaction time was measured and recorded automatically. Outliers (values outside of the limits of 3 standard deviations) have been automatically eliminated. The Stroop-Test is characterized by a high test-retest reliability.
  Due to the cross-over design of the study two days were necessary to determine the interventional effect. According to the group allocation the participants executed the Stroop-test either in an alternating or sitting posture. Differences in reaction time and accuracy between "alternating" and "sitting" days will be analyzed.
Attentional performance | 2 experimental days
  As the effect of alternating postures on attentional performance is still unclear, an attentional performance test called "d2R-test of attention" has been implemented. The d2R-test was executed as a pen and paper version. Therefore, it enabled screen breaks during the test protocol and simulated paper-related office work. The d2R-Test is characterized by a high test-retest reliability and do not require any specific previous knowledge except of rudimentary language skills. Normative values for the d2R-test are available for different countries.
  Attentional performance and accuracy were manually determined according to the d2R-guidelines.
  Due to the cross-over design of the study two days were necessary to determine the interventional effect. According to the group allocation the participants executed the d2R-test either in an alternating or sitting posture. Differences in attentional performance and accuracy between "alternating" and "sitting" days will be analyzed.
Working speed | 2 experimental days
  Physical efforts when performing standardized tests (e.g. standing or walking) can negatively influence cognitive parameters as well as working speed. To determine the effect of alternating postures on working speed a digital text editing task encouraging participants to fill in spaces in an ergonomic guideline text for 10 min was used.
  Working speed (words per minute) and accuracy (relative error) have been manually calculated.
  Due to the cross-over design of the study two days were necessary to determine the interventional effect. According to the group allocation the participants executed the text editing task either in an alternating or sitting posture. Differences in working speed between "alternating" and "sitting" days will be analyzed.
Workload perception | 2 experimental days
  Sit-to-stand workstations can evoke positive as well as negative associations. A common method to rate workload perception is the NASA-TLX questionnaire (Task Load Index, National Aeronautics and Space Administration). For reasons of simplicity and unmodified sensitivity, the short version of this questionnaire (RTLX, raw task load index), consisting of six major items, was used. Influences on workload perception based on unweighted items in the RTLX were negated due to the cross-over design.
  Due to the cross-over design of the study two days were necessary to determine the interventional effect. According to the group allocation the participants scored their perceived workload after executing several cognitive tests in an alternating or sitting posture. Differences in workload perception between "alternating" and "sitting" days will be analyzed.

OTHER OUTCOMES:
Body movements | 2 experimental days
  Body movements can alter physiological parameters and cognitive performance. Especially small movements during longer time intervals are very hard to classify by means of personal observations. Therefore, a three-dimensional accelerometer - placed on the sternum via a neoprene breast belt - was used to objectively measure body movements. Upper body placements of accelerometers have been shown to reliably detect body movements, and sit-to-stand as well as stand-to-sit transitions. To reduce the total number of sensors, a HRV-recorder with integrated 3D-accelerometer was used.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwartz, MSc, Study Director — University of Applied Sciences Upper Austria
Locations (1):
- University of Applied Sciences Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuhaus M, Healy GN, Dunstan DW, Owen N, Eakin EG. Workplace sitting and height-adjustable workstations: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):30-40. doi: 10.1016/j.amepre.2013.09.009. PMID 24355669
- [Background] Commissaris DA, Konemann R, Hiemstra-van Mastrigt S, Burford EM, Botter J, Douwes M, Ellegast RP. Effects of a standing and three dynamic workstations on computer task performance and cognitive function tests. Appl Ergon. 2014 Nov;45(6):1570-8. doi: 10.1016/j.apergo.2014.05.003. Epub 2014 Jun 17. PMID 24951234
- [Background] Bates ME, Lemay EP Jr. The d2 Test of attention: construct validity and extensions in scoring techniques. J Int Neuropsychol Soc. 2004 May;10(3):392-400. doi: 10.1017/S135561770410307X. PMID 15147597
- [Background] Best JR, Nagamatsu LS, Liu-Ambrose T. Improvements to executive function during exercise training predict maintenance of physical activity over the following year. Front Hum Neurosci. 2014 May 27;8:353. doi: 10.3389/fnhum.2014.00353. eCollection 2014. PMID 24904387
- [Background] Van der Elst W, Van Boxtel MP, Van Breukelen GJ, Jolles J. The Stroop color-word test: influence of age, sex, and education; and normative data for a large sample across the adult age range. Assessment. 2006 Mar;13(1):62-79. doi: 10.1177/1073191105283427. PMID 16443719
- [Background] Lynch BM. Sedentary behavior and cancer: a systematic review of the literature and proposed biological mechanisms. Cancer Epidemiol Biomarkers Prev. 2010 Nov;19(11):2691-709. doi: 10.1158/1055-9965.EPI-10-0815. Epub 2010 Sep 10. PMID 20833969
- [Background] Owen N, Sparling PB, Healy GN, Dunstan DW, Matthews CE. Sedentary behavior: emerging evidence for a new health risk. Mayo Clin Proc. 2010 Dec;85(12):1138-41. doi: 10.4065/mcp.2010.0444. No abstract available. PMID 21123641
- [Background] Brown WJ, Miller YD, Miller R. Sitting time and work patterns as indicators of overweight and obesity in Australian adults. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1340-6. doi: 10.1038/sj.ijo.0802426. PMID 14574344
- [Background] Schwartz B, Kapellusch JM, Schrempf A, Probst K, Haller M, Baca A. Effect of a novel two-desk sit-to-stand workplace (ACTIVE OFFICE) on sitting time, performance and physiological parameters: protocol for a randomized control trial. BMC Public Health. 2016 Jul 15;16:578. doi: 10.1186/s12889-016-3271-y. PMID 27422158
- [Derived] Schwartz B, Kapellusch JM, Schrempf A, Probst K, Haller M, Baca A. Effect of alternating postures on cognitive performance for healthy people performing sedentary work. Ergonomics. 2018 Jun;61(6):778-795. doi: 10.1080/00140139.2017.1417642. Epub 2017 Dec 28. PMID 29235967